CLINICAL TRIAL: NCT05173597
Title: The Performance of an Individual Dosing Regimen of Follitropin Delta for Controlled Ovarian Stimulation for IVF in a Real-word Setting: a Non-interventional Observational Study
Brief Title: Real-world Evidence on Follitropin Delta Individual Dosing
Status: Recruiting | Type: Observational
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. M.Sc. Georg Griesinger, Professor, University of Luebeck
Other Study IDs: Aktenzeichen 21-385
Record Dates: First submitted 2021-11-18; First posted 2021-12-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Infertility; Sterility
Keywords: In-Vitro-Fertilisation; Assisted reproduction; Ovarian Stimulation; Ovarian Hyperstimulation Syndrome
MeSH Terms: conditions — Infertility; Ovarian Hyperstimulation Syndrome | interventions — follitropin delta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving treatment with Follitropin-delta: The included patients are adult women from the routine clinical care settings with indication for ovarian stimulation with follitropin delta in a GnRH-antagonist protocol who are making a first treatment attempt IVF or ICSI. This study is intended to be conducted in non-vulnerable population. No vulnerable subjects will be enrolled in the study.
  Interventions: Drug: Follitropin delta

INTERVENTIONS:
Drug: Follitropin delta — REKOVELLE® (follitropin delta), solution for injection - delivered with an injection pen, ATC code G03GA10, is a recombinant human FSH approved for the controlled ovarian stimulation for the development of multiple follicles in women undergoing assisted reproductive technologies such as an in vitro fertilisation or intracytoplasmic sperm injection cycle.
  Other Names: REKOVELLE® (follitropin delta)

SUMMARY:
As part of the in vitro fertilisation treatment, ovarian stimulation is routinely performed. For this purpose, FSH preparations are used. Follitropin delta is a FSH preparation that is approved for a wide range of applications and is dosed individually according to body weight and serum anti-Müllerian hormone (AMH). Body weight is used to estimate the distribution volume of the glycoprotein FD in the patient and is thus a proxy of exposure. The AMH is used to estimate the ovarian reserve and thus the number of follicles in the ovaries that can be recruited by Follitropin delta stimulation. An algorithm is used for individual dosing. The aim of individual dosing is to reduce the probability of an under or overreaction of the ovaries to FSH therapy.

In contrast to phase III registration studies, patients with severe overweight and underweight, as well as very high and very low AMH values and associated disorders of the menstrual cycle and oocyte maturation, are also found in the reality of care. The performance of the dosing algorithm and thus the results of ovarian stimulation in these subgroups of patients have so far been insufficiently investigated in the phase III registration trials.

In the present study no statistical hypothesis will be tested. The study is descriptive by design and the analyses are descriptive and exploratory. NIS is chosen in order to explore how the individualized dosing regimen of REKOVELLE® performs in routine clinical practice and to investigate the effectiveness and safety of REKOVELLE® under real-world conditions. This is a monocentric, prospective, non-interventional cohort study conducted in normal care setting in a fertility clinic that will collect information from 850 women undergoing up to two cycles of IVF or ICSI treatment with controlled ovarian stimulation with REKOVELLE®.

DETAILED DESCRIPTION:
Infertility is often defined as the failure to achieve a pregnancy after 12 months or more of regular unprotected sexual intercourse. Many factors (age, gynaecological problems, life style factors) can cause infertility and may involve the male, the female or both.

Global estimates suggest that the 12-month prevalence rate of infertility ranged from 3.5% to 16.7% in developed countries, with a median prevalence of 9% worldwide for women aged 20 - 44 years. A recent study estimated that 1.9% of child-seeking women aged 20 - 44 years experienced primary infertility (unable to have a live birth) and 10.5% secondary infertility (at least one live birth). The proportion of infertile couples seeking any infertility medical care ranges from 51% in less developed countries to 56% in developed countries, and 22% actually received infertility treatment.

Among fertility treatment, controlled ovarian stimulation (COS) with recombinant or urinary follicle stimulating hormone (FSH) and human menotropin gonadotropin (hMG) aims to obtain an adequate number of competent oocytes to be used for assisted reproductive technologies (ART) such as an in vitro fertilisation (IVF) or intracytoplasmic sperm injection (ICSI), with minimum risks for the woman.

The ovarian response is influenced by the dose of gonadotropin, but there is a large variability across patients for the same dose of gonadotropin. A standard starting dose of gonadotropin in women with a low ovarian reserve may result in a poor ovarian response. In women with a high ovarian reserve, the same dose may result in an excessive response and therefore increases the risk of complications such as the ovarian hyperstimulation syndrome (OHSS). OHSS is a rare but critical complication associated with gonadotropin use. Severe OHSS occurs in approximately 1.4 % of all COS cycles.

Individualizing COS regimens is therefore crucial to ensure an appropriate dosing from the start of stimulation in order to reduce the risk of cycle cancellation due to poor response and minimize the iatrogenic risks due to an excessive response.The use of biomarkers, which can predict ovarian response to exogenous FSH stimulation, has been extensively investigated. Among the different biomarkers, the serum level of anti-müllerian hormone (AMH) is currently considered as the most robust marker of the ovarian reserve. In addition, AMH serum levels shows relative stability and consistency during the menstrual cycle, and can therefore be measured at any time of the menstrual cycle.

In December 2016, Ferring received Marketing Authorisation approval from the European Commission for follitropin delta (FE 999049) under the trade name REKOVELLE®, a new human recombinant FSH (rFSH). The indication is: "Controlled ovarian stimulation for the development of multiple follicles in women undergoing assisted reproductive technologies (ART) such as an in vitro fertilisation (IVF) or intracytoplasmic sperm injection (ICSI) cycle." This is the first rFSH treatment to be administered with an individualised dosing regimen, based on a woman's serum AMH level as well as her body weight.

This individualised dosing regimen was established in a phase-2 AMH-stratified trial conducted in 265 IVF/ICSI patients using pharmacokinetic (PK) and pharmacodynamic (PD) modelling and simulation. A robust assay was developed in collaboration with Roche Diagnostics to ensure a reliable assessment of AMH levels at the standards intended for companion diagnostics.

The efficacy and safety of Follitropin Delta was first evaluated in the ESTHER-1 (Evidence- based Stimulation Trial with Human rFSH in Europe and Rest of World) phase-3 trial, which compared the individualized Follitropin Delta dosing based on AMH level and body weight with conventional Follitropin Alfa (Gonal-F®) dosing. Patients who did not achieve an ongoing pregnancy could continue in the ESTHER-2 phase-3 trial, which evaluated the immunogenicity in repeated COS cycles. The results of the phase-3 trials showed that individualized Follitropin Delta was non-inferior to conventional Follitropin Alfa for ongoing pregnancy and ongoing implantationrates. Overall, women treated with individualized Follitropin Delta dosing reached more frequently the prespecified optimum oocyte yield (8-14 oocytes), with fewer cases of extreme ovarian responses, and a reduced need for OHSS preventive measures.

The phase III clinical program has demonstrated that REKOVELLE® is an effective and well-tolerated treatment for controlled ovarian stimulation. Nevertheless, while clinical trials provide crucial information about drug efficacy and safety under controlled conditions in a selected group of patients, broader information is needed to explore how the individualized dosing regimen of REKOVELLE® is used in routine clinical practice and to investigate the effectiveness and safety of REKOVELLE® under real-world conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 to ≤ 44 years at enrolment

  * Planned stimulation in a fixed or flexible GnRH antagonist protocol
  * Planned use of follitropin delta for ovarian stimulation as per SmPC
  * Planned IVF or ICSI treatment with ejaculated or cryopreserved male germ cells, autologous or heterologous, with or without planned genetic testing of the oocytes or embryos
  * Planned preservation of MII oocytes (fertility preservation)
  * Planned triggering of final oocyte maturation with hCG or a GnRH agonist
  * Willingness and consent to participate

Exclusion Criteria:

* Serum AMH within 12 months prior to treatment ≤0.3 ng/ml
* Most recent serum AMH value before start of stimulation older than 12 months
* Serum AMH value not determined in Roche Elecsys immunoassays
* Pre-treatment with a combined oral contraceptive "pill" consisting of ethinyl estradiol and a synthetic progestogen

Ages: 18 Years to 44 Years | Sex: All
Age Groups: Adult
Study Population: The included patients are adult women from the routine clinical care settings with indication for ovarian stimulation with follitropin delta in a GnRH-antagonist protocol who are making a first treatment attempt IVF or ICSI. This study is intended to be conducted in non-vulnerable population. No vulnerable subjects will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Ovarian response | 2021-2022
  Number of cumulus-oocyte-complexes of the individual dosing regimen of follitropin delta for controlled ovarian stimulation for in-vitro fertilisation (IVF) or intracytoplasmic sperm injection (ICSI) in a cohort of patients from a real-world setting with focus on high body weight.

SECONDARY OUTCOMES:
Overall treatment outcome | 2021-2022
  Incidence of live birth stratified for low, normal and high AMH and body weight
Change in body weight | 2021-2022
  Determine change in body weight between 1st and 2nd cycle in subjects undergoing two cycles
Incidence of dose changes | 2021-2022
  Incidence of dose changes between 1st and 2nd treatment cycle in subjects undergoing two cycles
Intra-individual variation of ovarian response | 2021-2022
  Intra-individual variation of the number of cumulus-oocyte-complexes retrieved between 1st and 2nd treatment cycle in subjects undergoing two cycles, stratified for low, normal and high AMH and body weight and cycle regularity
Measurement of correlation of variance of body weight and AMH | 2021-2022
  Correlation coefficient of variance of body weight and AMH with variance of ovarian response between 1st and 2nd cycle in subjects undergoing two cycles
Comparison of intra-individual variance | 2021-2022
  Intra-individual variance in the number of cumulus-oocyte-complexes retrieved between first and second cycle in subgroups on the prospectively collected data and historical controls
Safety of treatment | 2021-2022
  Incidence of adverse events related to treatment and assessed by CTCAE v4.0 of follitropin delta in a real-world setting
Change in AMH | 2021-2022
  Difference in serum AMH values between 1st and 2nd cycle in subjects undergoing two cycles

CONTACTS AND LOCATIONS:
Locations (1):
- University of Luebeck, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zegers-Hochschild F, Adamson GD, de Mouzon J, Ishihara O, Mansour R, Nygren K, Sullivan E, Vanderpoel S; International Committee for Monitoring Assisted Reproductive Technology; World Health Organization. International Committee for Monitoring Assisted Reproductive Technology (ICMART) and the World Health Organization (WHO) revised glossary of ART terminology, 2009. Fertil Steril. 2009 Nov;92(5):1520-4. doi: 10.1016/j.fertnstert.2009.09.009. Epub 2009 Oct 14. PMID 19828144
- [Background] Practice Committee of the American Society for Reproductive Medicine. Diagnostic evaluation of the infertile male: a committee opinion. Fertil Steril. 2015 Mar;103(3):e18-25. doi: 10.1016/j.fertnstert.2014.12.103. Epub 2015 Jan 15. PMID 25597249
- [Background] Practice Committee of American Society for Reproductive Medicine. Diagnostic evaluation of the infertile female: a committee opinion. Fertil Steril. 2012 Aug;98(2):302-7. doi: 10.1016/j.fertnstert.2012.05.032. Epub 2012 Jun 13. PMID 22698637
- [Background] Boivin J, Bunting L, Collins JA, Nygren KG. International estimates of infertility prevalence and treatment-seeking: potential need and demand for infertility medical care. Hum Reprod. 2007 Jun;22(6):1506-12. doi: 10.1093/humrep/dem046. Epub 2007 Mar 21. PMID 17376819
- [Background] Mascarenhas MN, Flaxman SR, Boerma T, Vanderpoel S, Stevens GA. National, regional, and global trends in infertility prevalence since 1990: a systematic analysis of 277 health surveys. PLoS Med. 2012;9(12):e1001356. doi: 10.1371/journal.pmed.1001356. Epub 2012 Dec 18. PMID 23271957
- [Background] Arce JC, Andersen AN, Fernandez-Sanchez M, Visnova H, Bosch E, Garcia-Velasco JA, Barri P, de Sutter P, Klein BM, Fauser BC. Ovarian response to recombinant human follicle-stimulating hormone: a randomized, antimullerian hormone-stratified, dose-response trial in women undergoing in vitro fertilization/intracytoplasmic sperm injection. Fertil Steril. 2014 Dec;102(6):1633-40.e5. doi: 10.1016/j.fertnstert.2014.08.013. Epub 2014 Sep 23. PMID 25256937
- [Background] Practice Committee of American Society for Reproductive Medicine. Ovarian hyperstimulation syndrome. Fertil Steril. 2008 Nov;90(5 Suppl):S188-93. doi: 10.1016/j.fertnstert.2008.08.034. PMID 19007627
- [Background] Kupka MS, Ferraretti AP, de Mouzon J, Erb K, D'Hooghe T, Castilla JA, Calhaz-Jorge C, De Geyter C, Goossens V; European IVF-Monitoring Consortium, for the European Society of Human Reproduction and Embryology. Assisted reproductive technology in Europe, 2010: results generated from European registers by ESHREdagger. Hum Reprod. 2014 Oct 10;29(10):2099-113. doi: 10.1093/humrep/deu175. Epub 2014 Jul 27. PMID 25069504
- [Background] Klemetti R, Sevon T, Gissler M, Hemminki E. Complications of IVF and ovulation induction. Hum Reprod. 2005 Dec;20(12):3293-300. doi: 10.1093/humrep/dei253. Epub 2005 Aug 26. PMID 16126753
- [Background] La Marca A, Sunkara SK. Individualization of controlled ovarian stimulation in IVF using ovarian reserve markers: from theory to practice. Hum Reprod Update. 2014 Jan-Feb;20(1):124-40. doi: 10.1093/humupd/dmt037. Epub 2013 Sep 29. PMID 24077980
- [Background] Broekmans FJ, Kwee J, Hendriks DJ, Mol BW, Lambalk CB. A systematic review of tests predicting ovarian reserve and IVF outcome. Hum Reprod Update. 2006 Nov-Dec;12(6):685-718. doi: 10.1093/humupd/dml034. Epub 2006 Aug 4. PMID 16891297
- [Background] Nelson SM. Biomarkers of ovarian response: current and future applications. Fertil Steril. 2013 Mar 15;99(4):963-9. doi: 10.1016/j.fertnstert.2012.11.051. Epub 2013 Jan 8. PMID 23312225
- [Background] La Marca A, Sighinolfi G, Radi D, Argento C, Baraldi E, Artenisio AC, Stabile G, Volpe A. Anti-Mullerian hormone (AMH) as a predictive marker in assisted reproductive technology (ART). Hum Reprod Update. 2010 Mar-Apr;16(2):113-30. doi: 10.1093/humupd/dmp036. Epub 2009 Sep 30. PMID 19793843
- [Background] Anckaert E, Smitz J, Schiettecatte J, Klein BM, Arce JC. The value of anti-Mullerian hormone measurement in the long GnRH agonist protocol: association with ovarian response and gonadotrophin-dose adjustments. Hum Reprod. 2012 Jun;27(6):1829-39. doi: 10.1093/humrep/des101. Epub 2012 Apr 3. PMID 22473395
- [Background] Broer SL, Broekmans FJ, Laven JS, Fauser BC. Anti-Mullerian hormone: ovarian reserve testing and its potential clinical implications. Hum Reprod Update. 2014 Sep-Oct;20(5):688-701. doi: 10.1093/humupd/dmu020. Epub 2014 May 12. PMID 24821925
- [Background] La Marca A, Stabile G, Artenisio AC, Volpe A. Serum anti-Mullerian hormone throughout the human menstrual cycle. Hum Reprod. 2006 Dec;21(12):3103-7. doi: 10.1093/humrep/del291. Epub 2006 Aug 21. PMID 16923748
- [Background] Gassner D, Jung R. First fully automated immunoassay for anti-Mullerian hormone. Clin Chem Lab Med. 2014 Aug;52(8):1143-52. doi: 10.1515/cclm-2014-0022. PMID 24622790
- [Background] Nyboe Andersen A, Nelson SM, Fauser BC, Garcia-Velasco JA, Klein BM, Arce JC; ESTHER-1 study group. Individualized versus conventional ovarian stimulation for in vitro fertilization: a multicenter, randomized, controlled, assessor-blinded, phase 3 noninferiority trial. Fertil Steril. 2017 Feb;107(2):387-396.e4. doi: 10.1016/j.fertnstert.2016.10.033. Epub 2016 Nov 29. PMID 27912901